CLINICAL TRIAL: NCT05187676
Title: Study of the Concordance Between Skin Oxygen Saturation Measurements Made by an Innovative Non-contact Optical Imaging Device (IPAM) and the Reference Medical Device (Periflux 6000) in Patients With Skin Vascular Disorders or Chronic Wounds
Brief Title: Clinical Evaluation of an Innovative Non-contact Optical Device for Skin Oxygenation Imaging
Acronym: IMOXY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A03140-39
Record Dates: First submitted 2021-06-29; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-06

CONDITIONS: Chronic Wounds; Obliterating Arteriopathy of the Lower Limbs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxygen cutaneous saturation rate (ScO2) then transcutaneous oxygen partial pressure (TcPO2) (Experimental): ScO2 values will be measured using IPAM first then TcPO2 values will be measured using Periflux6000. ALways in the same order.
  Interventions: Device: Oxygen saturation measurement using the IPAM device; Device: Transcutaneous oxygen partial pressure (TcPO2) using the PeriFlux6000 device

INTERVENTIONS:
Device: Oxygen saturation measurement using the IPAM device — Skin oxygen saturation rate will be measured (%) using the non-contact optical device under evaluation called IPAM
Device: Transcutaneous oxygen partial pressure (TcPO2) using the PeriFlux6000 device — Skin TcPO2 will be measured (mmHg) using the reference device called PeriFlux6000

SUMMARY:
According to international consensus, information on the level of skin oxygenation is necessary for the diagnostic management of chronic wounds. The measurement of transcutaneous partial oxygen pressure (or TcPO2, according to the acronym) is measurable with a medical device that uses a Clark electrode. Since the medical device in question is expensive and the measurement time-consuming (approximately 45 minutes per patient), the TcPO2 is only rarely accessible (in hospital medicine as in nursing homes) and is therefore not predominant in the clinical decision. The clinical decision is currently mainly based on the result of the ankle blood pressure measurement, which is readily available.

The main objective is to study, from the same skin surfaces (same localization of skin sites and same dimensions of each surface in cm²), in patients with cutaneous vascular disorders or chronic wounds, the relationship between (i) the transcutaneous oxygen saturation values (expressed as a percentage) by the innovative non-contact optical imaging device under study (IPAM, method to be validated) and (ii) the transcutaneous partial oxygen pressure values (TcPO2) (expressed in millimeters of mercury, mmHg) measured by the reference medical device (Périflux6000, gold standard).

DETAILED DESCRIPTION:
The InnovaTICs Dépendance project, funded by the Grand Region Is, aims to develop a medical device meeting the need to measure quickly and non-invasively the skin oxygen saturation. To do this, a device medical was developed by CRAN (Joint Research Unit of the University of Lorraine and CNRS); its industrial transfer was entrusted to the company SD Innovation to produce the VRPC device for "video-reconstruction of chronic wounds". The VRPC medical device makes it possible to measure skin oxygen saturation by an optical (atraumatic) and non-contact (non-invasive) method, more quickly than the current method proposes. The capacity of the VRPC device to measure in vivo variations in skin oxygen saturation was confirmed by carrying out measurements on healthy volunteers. The measured values made it possible to show that the VRPC device was able to detect the difference in skin oxygen saturation between the skin covering a "healthy" finger and the skin covering the same finger but after a tourniquet had been placed at the base of the first phalanx of the finger (data not published).

ELIGIBILITY:
Inclusion Criteria:

* Major,
* Having signed the informed consent to participate in the clinical study
* Compulsory affiliation to a social security scheme
* Presenting at least one of the following two criteria:

  * Presence of a PAD at the stage of Chronic Critical Ischemia (CHF) of stage III or IV according to the classification of Leriche and Fontaine,
  * Presence of one (or more) chronic wound (s) of the lower limbs of the pressure sore or ulcer type.

Exclusion Criteria:

* Person referred to in Articles L. 1121-5, L1121-6, L. 1121-7 and L1121-8 of the Public Health Code.
* Pregnant woman, parturient or nursing mother
* Minor (non-emancipated)
* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* Person of full age unable to express consent
* Persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric treatment under Articles L.3212-1 and L. 3213-1.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-03 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Linear regression between the skin oxygen saturation rate (ScO2) values and the Transcutaneous oxygen partial (TcPO2) pressure values | Through study completion, an average of 2 years
  The relationship between TcPO2 and ScO2 measurements will be modeled

SECONDARY OUTCOMES:
Rate of clinical decision influenced by the IPAM device | Through study completion, an average of 2 years
  Questionnaire about the impact of the IPAM measurement on the clinical decision
Variation coefficient of the IPAM measurement made 3 times in a row on 3 different skin sites | Through study completion, an average of 2 years
  Repeatability of the IPAM measurement made 3 times in a row on 3 different skin sites
Duration of use in seconds | Through study completion, an average of 2 years
  Comparison of the mean duration time for acquiring one measurement with each of the devices used in the study
Skin surface accessible for measurement in square centimeters | Through study completion, an average of 2 years
  Comparison of the mean skin surface on which skin oxygen saturation rate and TcPO2 may be measured by each of the two medical devices used fot his study
Ergonomics evaluation in terms of physical and mind efforts | Through study completion, an average of 2 years
  Using a scale already used for medical devices ergonomics evaluation, the ergonomics of the two devices will be compared
Mosaicing software success rate | Through study completion, an average of 2 years
  The mosaicing software will be evaluated on a 20s-duration video sequence
Risk evaluation: redness will be evaluated on a scale from zero to ten | Through study completion, an average of 2 years
  Skin reddening will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, Mills JL, Ricco JB, Suresh KR, Murad MH; GVG Writing Group. Global vascular guidelines on the management of chronic limb-threatening ischemia. J Vasc Surg. 2019 Jun;69(6S):3S-125S.e40. doi: 10.1016/j.jvs.2019.02.016. Epub 2019 May 28. PMID 31159978